CLINICAL TRIAL: NCT04787081
Title: Nighttime Postural Care: Caregiver Training Program and Outcome Measure Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Catherine University (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 938
Record Dates: First submitted 2021-01-22; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-01

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: competence post learning; nighttime postural care education; online caregiver education; postural care; cerebral palsy; sleep positioning
MeSH Terms: conditions — Behavior; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Mixed methods double-blind parallel group design, involving a consecutive sample of adults being randomly assigned to an educational intervention (Group A or B). The Principal Investigator enrolled participants, designating subject numbers and professional or non-professional labels. The research assistant completed randomization, drawing concealed numbers from an envelope to determine participant's educational intervention group (A or B). To balance the number of professionals and non-professionals across groups, the research assistant used co-variate adaptive group randomization and applied a difference threshold of 3.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators hypothesized that caregivers would be more competent after lesson A (as compared with lesson B). Because of this participants were masked from knowing which lesson they'd received and were not informed about investigators hypothesis. The clinician's responsible for measuring participants' observed competence for positioning a person post-training were not informed of participant's assigned lesson. Participants were instructed to not discuss their lesson or lesson details with the clinicians' measuring those outcomes. The research assistant completed randomization and academic technology personnel registered participants into their lesson to ensure the principal investigator was not informed of participant's assigned lesson.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Care Positioning Training Program GRP1 (Experimental): A sleep care positioning lesson created by a University's postural-care scholars using Camtasia® video creation software with modules on evidence for night-time postural care, risk factor monitoring, sleep system types and set up, positioning methods, and outcome measures. This lesson consisted of interactive videos embedded with learning checkpoints. All videos included narration and closed captioning. The following link contains the videos which were modified post-study to reflect some of the participant's feedback: https://stkatentpc.weebly.com/
  Interventions: Other: Sleep Care Positioning Training Program GRP1
- Sleep Care Positioning Training Program GRP2 (Active Comparator): A sleep care positioning lesson created by a research assistant along with the principal investigator with modules on evidence for night-time postural care, risk factor monitoring, sleep system types and set up, positioning methods, and outcome measures. This lesson consisted of primarily written summary statements and links to freely available web-based information. Most of this lesson's modules included written information that the participant would need to read with the exception of the positioning methods modules. For the positioning module, participants were provided with links to manufacturers' websites which contained video clips on how to place postural supports.
  Interventions: Other: Sleep Care Positioning Training Program GRP2

INTERVENTIONS:
Other: Sleep Care Positioning Training Program GRP1 — Video-based tutorial covering six nighttime postural care topic areas which contained narration and closed captioning. This 2-hour online training program was delivered in a University classroom via D2L Brightspace.
  Other Names: Lesson A
  Arms: Sleep Care Positioning Training Program GRP1
Other: Sleep Care Positioning Training Program GRP2 — Web-link based tutorial covering six nighttime postural care topic areas which contained mostly written content. This self-paced online training program was delivered in a University classroom via D2L Brightspace.
  Other Names: Lesson B
  Arms: Sleep Care Positioning Training Program GRP2

SUMMARY:
This experimental study investigated the feasibility of a sleep care positioning training protocol by comparing two educational interventions using a randomized control design. The overarching Population Intervention Comparison Outcomes (PICO) question was: Is the training protocol feasible for use in training caregivers? Question one includes the following sub questions: A. Is there a difference in perceived competence to implement aspects of nighttime postural care intervention or observed ability to position the person in a sleep system between caregivers receiving one training program versus another? B. Does the training protocol prepare caregivers to implement nighttime postural care (NTPC).

DETAILED DESCRIPTION:
Target Population

Investigators planned to recruit a convenience sample of 40 adult participants identified as professional or non-professional care providers (primarily from two community organizations that specialize in serving clients with CP). Care providers of children (aged 6-12) with severe CP (those with limited ability to move and/or whom require use of a wheelchair) were the primary target population, since this matches the intended sample of a future intervention study. However caregivers of children outside of the 6-12 age range whom were candidates for NTPC and had similar mobility limitations as those with severe CP would not be excluded. Professional care providers could be nurses, occupational and physical therapists, assistive technology providers, etc. Non-professional care providers could be family members, care attendants, etc. Only individuals with knowledge of the child's sleep habits or routines were to be included in the study

Investigators used a mixed methods double-blind parallel group design, randomly assigning a consecutive sample of adults to an educational intervention (Lesson A or Lesson B).

Participant Recruitment

Investigators emailed flyers, recruiting participants from clinics serving persons with CP and universities educating healthcare providers and included professional and non-professional caregivers of persons with movement disorders, primarily CP with knowledge of a child's sleep habits and routines.

Participant activities

Participants completed study activities on one scheduled date: Consent process, baseline questionnaire (immediately before training), online education, post-training questionnaire, positioning of a simulated "client", post-simulation questionnaire, and exit interview. Participants completing all aspects of the study received a $50 gift card.

Randomization and blinding

The Principal Investigator (PI) enrolled participants, designating subject numbers and professional or non-professional labels. The research assistant completed randomization, drawing concealed numbers from an envelope, using Zelen's model of co-variate adaptive group randomization, and applying a threshold difference of three to balance professionals and non-professionals. An information technologist registered participants into their assigned lesson. At most five participants at a time were allowed in a classroom, with each room assigned a single lesson (A or B). Research assistants instructed participants on accessing and navigating their lesson and keeping details confidential. These processes helped ensure the PI, participants, and clinician simulation raters were not informed of lesson assignment.

Participants had the option to complete the non-assigned lesson in addition to their assigned lesson. Investigators verified participants' completion of all research activities (besides the exit interview) before the optional non-assigned lesson.

Intervention similarities and differences

Both online lessons included modules on evidence for NTPC, risk factor monitoring, sleep system types and set up, positioning methods, and outcome measures and were delivered via D2L Brightspace, a cloud-based learning management system. Both lessons' positioning-methods modules included video-based instruction. Lesson formats differed by source and design: Lesson A, created by a university's postural-care scholars using Camtasia® video creation software, consisted of interactive videos embedded with learning checkpoints, while Lesson B included written summary statements and links to freely available web-based information.

Simulation

Following their lesson and post-training questionnaire, participants positioned a "client" in a hospital bed using a designated commercial sleep system (henceforth termed "simulation"). The investigators followed protocols, instructing that participants position the client to the best of their ability, not using notes or asking observers for help; the "client" be positioned using straps to facilitate tight hamstrings in an asymmetrical-lying position common for persons with CP (i.e. head turned left, legs windswept right and knee flexed); and the clinician raters should complete the room set-up with the bed centered against the north wall, sleep system parts arranged consistently on a designated table, and that they should sit at predetermined observational locations.

Simulation raters

Health practitioners (two at a time) serving as clinician raters used the simulation observation instrument, independently observing and documenting a participant's positioning skills. An assistive technology professional and occupational therapist served as primary raters, rating 30 and 29 participants, respectively. Two secondary raters (both occupational therapists, one the PI) completed the remaining observations.

Data collection measures

Investigators collected quantitative and qualitative data using questionnaires for obtaining participants' self-perceptions of competence and lesson feedback. An observation instrument was used for scoring and describing participants' simulation performance. Fieldnotes were used for recording participant activities across the study period. The PI designed all study instruments, after reviewing competency literature, conducting a pilot study (unpublished) and consulting an academic measurement expert.

Statistical power

Before data collection, investigators chose a significance level (0.05) with plans for enrolling a minimum of 30 participants. With 15 participants per group, so there would be 80% power to detect a difference between groups of 1.06 standard deviations, where "standard deviation" describes variation within groups (i.e., Cohen's d = 1.06). Because this is the first study examining caregivers' NTPC competence from online education, no prior data could inform power calculation or supply a "standard deviation" value.

Data analysis, quantitative outcomes

Perceived Competence. Each participant provided a total average perceived competence score (total average from knowledge, ability and confidence sub-scores) at three times: baseline, post-training, and post-simulation. Investigators analyzed these scores using a mixed linear model; the random effect was participant, and fixed effects were group (Lesson A or Lesson B), professional vs. non-professional status, time (baseline, post-training, and post-simulation), and all two-way and three-way interactions. Investigators tested change over time within groups using a contrast in the group-by-time interaction (which combines professionals and non-professionals) and compared groups at each time also using contrasts in the group-by-time interaction. Statistical analyses used JMP (v. 14.0.0 Pro, SAS Institute, Cary NC).

Observed competence. Investigators computed participants' average positioning/simulation score (number correct out of 16 tasks from the simulation observation instrument) and used a mixed linear model to examine differences in observed positioning ability based on group (Lesson A or B) and professional vs. non-professional status.

Correlation of perceived and observed competence. Investigators used Pearson's correlation (r) to measure the association between participants' average self-ratings on positioning-based competence items and their average correct positioning/simulation scores, to understand the groups' ability to self-assess performance.

Interrater Reliability. Investigators measured interrater reliability using the intra-class correlation (ICC), once including all simulation observation raters and separately including the two primary clinician raters and the PI.

Data analysis, qualitative

For qualitative data, investigators used a modified grounded theory approach of open, axial and selective coding similar to that described by Bhattacherjee. From questionnaire and exit interview data, the PI read line-by-line, coding responses into categories and themes. From the simulation observation instrument, the PI listed each participant's incorrectly completed tasks and used a table to organize those tasks most frequently missed or completed incorrectly. Then clinicians' descriptive statements corresponding to incorrectly completed tasks were tabulated and reviewed line-by-line and coded into categories and themes.

Note: In addition to the above stated plan for examining the feasibility of the sleep care positioning training program, investigators also planned to examine the internal consistency reliability of the sleep disturbance scale for children (SDSC), a 27-item inventory rated on a 5 point Likert-type scale which was created by Bruni et al in 1996. To examine its reliability, study participants who self-identified as having night to night knowledge of a child with cerebral palsy's sleep performance were asked to complete the SDSC. While data was collected for this aspect of the study, only 10 participants self-identified as having such knowledge; thus, further analysis of the tools' reliability was not completed by investigators.

ELIGIBILITY:
Inclusion Criteria:

* Professional and non-professional caregivers of children with movement disorders or cerebral palsy.

Exclusion Criteria:

* Caregivers without knowledge of sleep habits and routines of persons with such diagnoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-22 (Actual); Study Completion 2018-09-22 (Actual)

PRIMARY OUTCOMES:
Baseline Sleep Care Positioning Questionnaire | Completed immediately before training/educational intervention. Same day as training.
  Perceived competence questionnaire with 4-pt. ratings of knowledge, ability and confidence for nighttime postural care research, risk factor monitoring, sleep system types / set-up, positioning a person, and measuring outcomes.
Post Sleep Care Positioning Program Questionnaire | Completed immediately after training / educational intervention. Same day as training.
  Perceived competence questionnaire with 4-pt. ratings of knowledge, ability and confidence for nighttime postural care research, risk factor monitoring, sleep system types / set-up, positioning a person, and measuring outcomes.
Post Simulation Sleep Care Positioning Program Questionnaire | Completed immediately after simulation activity, after positioning a person in a sleep system. Same day as training.
  Perceived competence questionnaire with 4-pt. ratings of knowledge, ability and confidence for nighttime postural care research, risk factor monitoring, sleep system types / set-up, positioning a person, and measuring outcomes.

SECONDARY OUTCOMES:
Simulation Observation Instrument | Completed after training and post-training questionnaire. Same day as training.
  Instrument with list of 16 positioning tasks with Yes/No columns meant for raters to check for each task, indicating whether or not task was completed by participant. Additionally this instrument included space and directions for raters to record observations of participants from the start to end of the simulation/positioning the person activity.

CONTACTS AND LOCATIONS:
Overall Officials: John Schmitt, Study Chair — St. Catherine University
Locations (1):
- St. Catherine University, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing plan will be determined based on researcher requests. The following could potentially be shared: blank informed consent document (attached to this registry), protocol submitted to IRB (attached to this registry), blank questionnaires and simulation observation instruments and de-identified raw numerical data from questionnaire and simulation observation instrument.
Supporting Information: Study Protocol, ICF
Time Frame: January, 2021 - January 2022
Access Criteria: Please email any requests for additional information to Jennifer Hutson at jahutson@stkate.edu

REFERENCES:
- [Background] Hutson, J.A. (2020). Nighttime Postural Care Sleep-Based Outcome Measures and Education: Preparing Care Providers of Children with Cerebral Palsy (Doctoral Dissertation). University of Minnesota, Available from ProQuest Dissertations Publishing. (Dissertation Number: 27741484)
- See also: The sleep care positioning training program (Lesson A) which was provided to Group 1. The version found at this site contains some edits based on the feedback provided by participants during the research study. — https://stkatentpc.weebly.com/
- See also: Jennifer Hutson's dissertation which contains a detailed description of the study and its outcomes (information about this study is primarily contained within chapters 3 & 4 of the dissertation). — https://works.bepress.com/jennifer-hutson/11/

DOCUMENTS (2):
  • Informed Consent Form (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT04787081/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-04-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT04787081/Prot_SAP_001.pdf